CLINICAL TRIAL: NCT00906659
Title: Correlation of Visual Function, Center Point Thickness and Macular Volume Changes Three Weeks After Focal Photocoagulation for Diabetic Macular Edema
Brief Title: Visual Function, Center Point Thickness and Macular Volume After Photocoagulation
Status: Completed | Type: Observational
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Virgilio Lima Gomez, Hospital Juarez de Mexico
Other Study IDs: HJM 1453/08.02.26
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Diabetic Retinopathy; Macular Edema
Keywords: center point thickness; diabetic retinopathy; diabetic macular edema; macular volume; visual capacity; visual function
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetic macular edema: type 2 patients who had been treated with selective photocoagulation for clinically significant macular edema

SUMMARY:
The purpose of this study is to correlate changes of visual function three weeks after photocoagulation for macular edema, with changes of center point thickness and macular volume.

DETAILED DESCRIPTION:
Photocoagulation for clinically significant macular edema is effective to reduce the incidence of moderate visual loss. Selective photocoagulation for focal macular edema statistically reduces macular thickening, measured with optical coherence tomography, as early as two weeks after treatment, without significant changes over center point thickness. Although anatomic improvement has been demonstrated with OCT, clinical improvement takes longer to be evident: the Early Treatment Diabetic Retinopathy Study describe that clinical differences in visual function are after the eight month, and all the treatment strategies for macular edema used in this study were associated with an increased rate of moderate visual loss, during the first six weeks. Differences in research can achieve statistical significance, without clinical significance. A study was conducted to identify changes of visual function three weeks after photocoagulation for focal macular edema, and to correlate them with changes of CPT and macular volume, in order to compare the behavior of anatomical changes with visual changes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* regardless of diabetes duration and retinopathy severity level
* one or both eyes with focal clinically significant macular edema
* treated with selective or focal photocoagulation
* visual capacity under subjective refraction before and three weeks after treatment
* adequate quality 6 mm fast macular map both on the day of photocoagulation, and three weeks after it

Exclusion Criteria:

* patients with myopia over -6.00 diopters
* any retinal disease different from diabetic retinopathy at the moment of photocoagulation
* eyes with a thickened posterior vitreous
* eyes with vitreoretinal traction at the macula
* if they had required scatter photocoagulation before the three weeks evaluation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population were type 2 diabetics from Mexico City and its metropolitan area, accessible population were the patients who attended a General Hospital in Mexico City
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
visual capacity (under subjective refractive correction was measured in decimal equivalent) | before the treatment and 3 weeks after photocoagulation
center point thickness (measured in µm) | before the treatment and 3 weeks after photocoagulation
macular volume (measured in mm3) | before the treatment and 3 weeks after photocoagulation

CONTACTS AND LOCATIONS:
Overall Officials: Dulce M Razo Blanco Hernandez, MD, Study Director — Hospital Juarez de Mexico; Virgilio Lima Gomez, MD, MSc, Study Chair — Hospital Juarez de Mexico; Aleyda S Cruz Diaz, MD, Principal Investigator — Hospital Juarez de Mexico
Locations (1):
- Hospital Juarez de Mexico, Mexico City, Mexico City, Mexico